CLINICAL TRIAL: NCT06028659
Title: Investigation of in Vivo Endogenous and/or Exogenous Production of Phenolic Metabolites Using (un)Targeted Metabolomics
Acronym: ENDOPHENOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Pedro M. Mena Parreño, Principal Investigator, University of Parma
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: 340/2023/SPER/UNIPR
Record Dates: First submitted 2023-08-23; First posted 2023-09-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-01

CONDITIONS: Individual Variability in (Poly)Phenol Metabolism
Keywords: (poly)phenols; catabolites; coffee; metabolism; low-molecular-weight (poly)phenols; metabolomics
MeSH Terms: interventions — Coffee; Water

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coffee (Experimental): In this arm, volunteers will receive, once, 3 decaffeinated coffees (150 mL total) with sugar as a known source of (poly)phenols.
  Interventions: Other: Coffee
- Control (Other): In this arm, volunteers will receive, once, 150 mL of sugared water as control.
  Interventions: Other: Water

INTERVENTIONS:
Other: Coffee — Decaffeinated coffee with 1 pack (5g) of sugar from commercially available brands prepared with commercially available domestic coffee machines.
  Arms: Coffee
Other: Water — 150 mL of hot water with 1 pack (5g) of sugar from commercially available brands prepared with commercially available domestic coffee machines.
  Arms: Control

SUMMARY:
Plant (poly)phenols is what we call a large number of substances that are produced by plants as secondary plant metabolites, which means substances that are not used for their growth and development but are necessary for them to survive. (Poly)phenols are divided in two major groups, flavonoids, and non-flavonoids, and each group contains a varied set of subgroups and substances. They are widely spread in fruit and vegetables that are part of the human diet, and, in general, studies have attributed many biological effects to the ingestion of (poly)phenols, especially in the prevention of non-communicable diseases. For this reason, research aims to understand their role in the health benefits of a diet that is rich in fruits and vegetables. When ingested, (poly)phenols are digested by both the human organism and the gut microbiota and are broken down into several smaller substances (catabolites) that are called low-molecular weight (poly)phenols (LMWP). Most of the absorbed (poly)phenols that reach our bloodstream and organs are LMWP.

For the proposed study, 30 healthy adults will be recruited and, if considered able to participate, will follow a standardized diet that is restricted in (poly)phenol intake and will be randomly divided into two groups: one will receive a known source of (poly)phenols (coffee) and the other will receive water, keeping the restriction of (poly)phenol from the diet. The duration of one phase is 4 days + 12 hours, during which urine, feces, and saliva will be collected. Then, after a 2-week-interval, subjects will repeat the experiment, except that this time the group who had coffee will have water, and vice versa. Again, urine and feces will be collected. The objective of the study is to identify and quantify LMWP mainly in urine, but also in feces, and try to understand how much was produced when there was no (poly)phenols in the diet compared with when there was ingestion of coffee (poly)phenols. The production of LMWP without coffee could be because of their production from other sources, like the metabolism of amino acids, proteins, and catecholamines (i.e. dopamine). The composition of the gut microbiota and relevant genetic information can alter the metabolism of (poly)phenols and will be considered in the analyses. Knowing how much of LMWP actually comes from the diet is important to understand the relevance and health benefits of these molecules.

DETAILED DESCRIPTION:
The study will consist of a randomized cross-over trial and each arm will last 5 days. A total of thirty (30) healthy volunteers will be recruited for the study in Parma (PR), using announcements placed in the university, hospital, and public places. To allocate subjects to each arm, a list will be generated using a randomized block design by using Random Number Generator Pro (Segobit Software). This list will be blind for the PI and volunteers, as it will be made by a colleague not involved in the subjects' enrolment and using a numbered sequence in sealed, opaque envelopes.

Volunteers freely accepting to participate to the study will be asked for their written informed consent. Information to the volunteers will be provided before and separately from the consent form. These information sheets and the informed consent forms have been prepared according to the Oviedo Convention and consider the guide of the local Ethics Committee. After obtaining their written informed consent, volunteers will undergo a screening visit to determine eligibility and collect personal data.

Privacy of the volunteers will be assured through pseudoanonymization by the attribution of a personal alphanumeric code. Recruited volunteers will also sign an authorisation to the use of personal information and retrieved data.

After recruitment, subjects will attend a first visit, when personal data will be collected, and body composition and anthropometry parameters measured. Then, they will receive the foods, supplements, and materials necessary to follow the study. The recruited subjects will be requested to follow a low-(poly)phenol diet, which will be the same for all the volunteers and maintained for the whole period of the intervention study. The foods, preparation mode, and times for eating the meals will be provided by the sponsor. The diet will be personalised to approximate the necessary calories based on the measured basal metabolic rate, multiplied by the physical activity level set at 1.45, and there will be quantitative variations on the low-(poly)phenol diet based on the daily energy requirement: 1500 kcal/day, 1750 kcal/day, 2000 kcal/day, 2250 kcal/day, 2500 kcal/day, 2750 kcal/day, or 3000 kcal/day, all with nutritionally balanced amounts of protein, fat, and carbohydrates. In addition, participants will be requested to restrict physical exercise during the study duration.

Subjects will be asked to collect urine produced during the 60h prior the intervention, starting from the evening prior the first day of diet (from 21.00 of the night prior the first day of diet) and every 12 hours (60-48h, 48-36h, 36-24h, 24-12h, 12-0h), and to complete the food diary to check for compliance to the diet. Subjects are asked to bring collected urine to the the Human Nutrition Unit of the Food and Drug Department of the University of Parma.

On the morning of the third day of diet, subjects will be requested to arrive at Parma University in fasting conditions. Prior to receiving the intervention, fasting spot urine and saliva samples will be collected. Then, sugared-decaffeinated-coffee (3 doses of 50 mL each and 5g of sugar) or sugared-water (150 mL of water and 5g of sugar) will be provided according to randomization of the arms, along with a standardized breakfast consisting of a (poly)phenol-free, nutritionally balanced solid meal and water (ad libitum).

After breakfast, subjects will be asked to autonomously collect urine for the next 48h at specified timepoints (0 - 3h; 3 - 6h; 6 - 9h; 9 - 12h; 12 - 24h; 24 - 36h; and 36 - 48h), following the same personalized diet. Lastly, subjects will autonomously collect a fecal sample within 6 to 48h after the intervention.

On the morning of the last day, after the last urine collection, subjects will bring collected urine and fecal samples and the 5-day food diary to the Human Nutrition Unit of the Food and Drug Department of the University of Parma.

After the first arm, subjects will resume their habitual lifestyles for 2 consecutive weeks, subsequently, they will attend another visit, when all the anthropometric evaluations carried out during the first visit will be repeated and another kit with foods and information for the personalized diet will be given. With the study being a cross-over design, the protocol followed will be the same as the one described above (except for saliva sampling, which will only be performed once). Coming the third day of diet, subjects who ingested coffee in the prior arm of the study will ingest water, and vice-versa.

For this study, the sample size was estimated considering the mean concentration of coffee-derived (poly)phenols and their metabolites in urine as the primary outcome and the available literature on similar approaches and studies of the area. The number of 30 volunteers was established considering the accepted parameters for clinical trials (power set at 0.8 and α set at 0.05) possible dropouts (15% drop-out rate), and exclusion of volunteers to maintain the sample power for statistical analysis. Before any comparison is performed, the normality of each variable will be evaluated to choose the most appropriate statistical test. If metabolite data are normally distributed, data will be expressed as mean ± standard deviation and analysed using repeated measures t-test or ANOVA with post-hoc comparisons. If data are not normally distributed, they will be reported as median and Interquartile Range and the Friedman test with post hoc pairwise comparisons will be performed. P-value < 0.05 will be regarded as statistically significant.

Unsupervised and supervised multivariate analysis will be used to identify and characterize the different urinary metabotypes, following the procedures developed by our research group for targeted metabolomics analysis of phenolic metabolites or when using untargeted metabolomics data. We will be using different clustering approaches to better explore the existing variability. This will serve to establish the number of clusters (i.e., phenolic metabotypes), the number of participants forming each cluster and the similarities among possible metabotypes.

The relationship between patterns of LMWP and their putative determinants (age, sex, ethnicity, lifestyle, anthropometrics, body composition, genotype, and gut microbiome) will be explored using correlation tests and multivariate analyses. P-value < 0.05 will be regarded as statistically significant. Statistics will be carried out by the specialized staff of the Human Nutrition Unit, under the supervision of the PI, and in collaboration with the University teams in charge of microbial profiling and genotyping.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy adults,
* Age 20-40 years old,
* Body mass index (BMI) between 18-28,
* Regular coffee consumers (at least 1 cup a day).

Exclusion Criteria:

* Clinical diagnosis of metabolic diseases,
* Clinical diagnosis of cardiovascular diseases,
* Clinical diagnosis of renal diseases,
* Clinical diagnosis of digestive diseases,
* Immunodeficiency
* Autoimmune diseases (other than well-compensated hypothyroidism),
* Mental disorders
* Regular use of medication (except birth-control pills and hormone replacement therapies),
* Use of antibiotics in the last month prior to enrollment,
* Food allergies or intolerances,
* Pregnancy
* Lactation

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number and concentration of phenolic metabolites in urine | Samples acquired from 60 hours prior to 48 hours after intervention or control
  Urine samples will be subjected to both targeted and untargeted liquid chromatography mass spectrometry analyses

SECONDARY OUTCOMES:
Identification and quantification of gut bacteria (genera and species) in feces | Samples acquired from 6-48 hours after coffee or control
  Analysis of microbiota taxonomy at species level from bacterial DNA extracted from fecal samples.
Number and concentration of phenolic metabolites in feces | Samples acquired from 6-48 hours after coffee or control
  Fecal samples will be subjected to both targeted and untargeted liquid chromatography mass spectrometry analyses
Identification and quantification of metabolites after in vitro fecal fermentation | Samples acquired from 6-48 hours after coffee or control
  A set of (poly)phenol-rich substrates and protein-rich food items will be incubated and fermented in sealed jars to evaluate the ability of human microbiota to produce different phenolic metabolites.
Identification of single-nucleotide polymorphism analysis | Single saliva samples collected from 1 hour to 30 minutes before the intervention with coffee or control.
  Genotyping for possibile genetic variations in genes related to (poly)phenol kinetics. Commercially available SNP arrays detect gene variability across the majority of the genome using a tagging SNP approach.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro M Mena Parreño, PhD, Principal Investigator — University of Parma
Locations (1):
- University of Parma - Plesso Biotecnologico Integrato, Parma, PR, Italy

IPD SHARING:
Plan to Share IPD: Yes
The data shared will be those that underlie results in a publication.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available from when published in peer-reviewed journals.
Access Criteria: Data available in publications can be freely accessed. If further data is required to be shared, it will be assessed case by case.

REFERENCES:
- [Derived] Zeraik L, Rosi A, Del Rio D, Crozier A, Bresciani L, Mena P. Endogenous and/or exogenous origin of phenolic metabolites in humans (the ENDOPHENOL project): study protocol for a randomized, controlled, crossover trial. Trials. 2025 Dec 19;26(1):571. doi: 10.1186/s13063-025-09215-9. PMID 41420184